CLINICAL TRIAL: NCT01789996
Title: Alternative Instruction in Six Minute Walk Test (6MWT)
Brief Title: The Six Minute Walk Test: Influence of Instruction on Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 10.089
Record Dates: First submitted 2013-02-09; First posted 2013-02-12 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2017-08

CONDITIONS: Interstitial Lung Disease
Keywords: 6 minute walk test; idiopathic pulmonary fibrosis; pulmonary arterial hypertension
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Pulmonary Arterial Hypertension | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternative six minute walk test (Active Comparator): Subjects will be given the following instructions
  1. walk as fast as they can in 6 minutes
  2. walk as normally as they can in 6 minutes
  3. walk leisurely as they can in 6 minutes. Pts will serve as their own controls.
  Interventions: Procedure: alternative six minute walk test
- Standard six minute walk test (Placebo Comparator): Subjects will be given the following instruction
  1. walk as far as they can in 6 minutes
  Interventions: Procedure: Standard six minute walk test

INTERVENTIONS:
Procedure: alternative six minute walk test — Alternate instructions will be given Subjects will
  1. walk as fast as they can in 6 minutes
  2. walk as normally as they can in 6 minutes
  3. walk leisurely as they can in 6 minutes. Pts will serve as their own controls.
  Other Names: fast vs far
  Arms: Alternative six minute walk test
Procedure: Standard six minute walk test — Subjects will walk as far as they can in 6 minutes
  Other Names: far
  Arms: Standard six minute walk test

SUMMARY:
Two - four 6MWT performed according to ATS standards. Each walk however had specifically altered wording and coaching performed in random order to determine differences in outcomes. One walk was done in the standard ATS fashion. One was done coaching to walk as fast as the patient can walk. One was coached to walk at the patients normal walking pace. One was coached to walk at the patient's leisure walking pace.

DETAILED DESCRIPTION:
Alternate 6MWT where subjects will be asked to walk as fast as they can, walk as normal as they can and walk leisurely as they can in 6 minutes compared to standard of care 6MWT which is walk as far as you can in 6 minutes.

ELIGIBILITY:
Inclusion Criteria:

* advanced lung disease such as COPD, ILD, IPF, or PAH

Exclusion Criteria:

* inability to walk, requiring supplemental oxygen, cardiac disease preventing successful 6MWT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
distance meters | 1 day
  this is an ongoing study of same day testing of 2-4 six minute walk tests, each with different instructions, to determine the impact of alternative instruction on outcome of the test

SECONDARY OUTCOMES:
oxygen saturation | 1 day
  assessed as an outcome of variable instruction given in different six minute walk tests performed in random order on the same day
dyspnea score | 1 day
  assessed as an outcome of variable instruction given in different six minute
heart rate response | 1 day
  assessed as an outcome of variable instruction given in different six minute

OTHER OUTCOMES:
heart rate recovery at one minute | 1 day
  assessed as an outcome of variable instruction given in different six minute

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Nathan, MD, Study Director — Inova Advanced Lung Disease and Transplant Program
Locations (1):
- Inova Advanced Lung Disease and Transplant Program, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We found that when the instruction was given to walk as fast as they can in six minutes, the distance was statistically greater than when the instruction was to walk as far as they can in six minutes. THe other instructions given yielded no difference in outcome. Other measures such are heart rate, Borg dyspnea score and saturation were not as statistically significant.

REFERENCES:
- [Derived] Weir NA, Brown AW, Shlobin OA, Smith MA, Reffett T, Battle E, Ahmad S, Nathan SD. The influence of alternative instruction on 6-min walk test distance. Chest. 2013 Dec;144(6):1900-1905. doi: 10.1378/chest.13-0287. PMID 23975232